CLINICAL TRIAL: NCT01748760
Title: Coping Long Term With Attempted Suicide - Adolescents
Acronym: CLASP-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Butler Hospital (Other)
Responsible Party: Principal Investigator, Shirley Yen, Assistant Professor (Research), Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH090147 (NIH)
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Results first posted 2017-01-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-09

CONDITIONS: Suicide
Keywords: Suicide Attempts; Suicidal Ideation
MeSH Terms: conditions — Suicide; Suicide, Attempted; Suicidal Ideation | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CLASP-A intervention (Experimental): Adolescent participants and parents will receive adjunctive psychosocial intervention.
  Interventions: Behavioral: CLASP-A intervention
- Treatment as Usual (Active Comparator): Adolescent participants and parents will not receive study intervention
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: CLASP-A intervention — Three individual sessions with adolescent patient using acceptance based strategies and motivational interviewing techniques. Sessions focused on identifying personalized risk factors for suicidal behavior, identifying values and goals, and development of personalized safety plan.
  Arms: CLASP-A intervention
Other: Treatment as Usual — Referral to outpatient treatment as part of routine discharge planning.
  Arms: Treatment as Usual

SUMMARY:
This study is to develop an adjunctive intervention for acutely suicidal adolescents who have been admitted to a psychiatric inpatient unit. The study intervention is comprised of: 1) two to three individual sessions delivered in an inpatient setting or immediately upon discharge; 2) one family session; 3) six months of follow-up phone interventions. The investigators hypothesize that those who receive the study intervention will have lower rates of suicide events and greater decreases in suicidal ideation after six months.

DETAILED DESCRIPTION:
The purpose of this R34 treatment development grant is to develop the "Coping Long-term with Attempted Suicide Program - Adolescents (CLASP-A)," an integrated, adjunctive intervention program for adolescents who have made a previous suicide attempt. The goals of CLASP-A are to reduce continued suicidal behavior and ideation, reduce risk behaviors for suicide, and improve adherence to psychosocial and psychopharmacologic treatments. It is comprised of three major components: a) three individual meetings while the patient is in the hospital, b) one in-person meeting with the patient and his/her parent/guardian in the hospital and c) a series of scheduled telephone contacts with the patient and parent/guardian for six months following discharge from the hospital. CLASP-A is based on a risk reduction model, and specifically targets four generic and potentially modifiable risk factors: hopelessness, impaired family support, problem solving deficits, and treatment non-adherence. The overall aim of this proposal is to further develop the CLASP-A intervention to address the needs of adolescents and to examine the feasibility and acceptability of this intervention program in adolescents. More specifically:

The development aims of this R34 proposal are to:

1. Develop CLASP-A - a multi-modal intervention that integrates strategies from cognitive-behavioral and values-based psychotherapies and family interventions, for use with suicidal adolescents.
2. Develop and implement adherence and competence rating scales to evaluate provider adherence to the intervention manual and their competence in delivering the intervention.
3. Improve the clarity, structure, content, acceptability, and feasibility of the intervention using information gathered from a small open trial (n=20) of adolescents, ages 12-18, who have made a recent suicide attempt.

The pilot study aims of this R34 proposal are to:

1. Conduct a randomized controlled pilot study in a sample of adolescent inpatients (n=50), ages 12-18, with a recent suicide attempt to assess the feasibility and acceptability of the proposed intervention and the randomization process.
2. To examine in an exploratory manner, preliminary evidence for the following hypotheses. It is expected that over a 6 month intervention period, compared to an enhanced treatment as usual (E-TAU) condition, adolescents assigned to CLASP-A + ETAU will have:

   1. fewer suicidal events, operationalized as a dichotomous composite score of suicide attempts, emergency department visits and inpatient hospital admissions due to suicide risk, and study rescue procedures due to suicide risk;
   2. lower suicidal ideation and less chronic suicidal ideation;
3. To examine in exploratory analyses potential mechanisms of change including treatment adherence to other forms of treatment as well as improvement in the hypothesized risk factors (i.e., hopelessness, problem-solving, and family functioning) addressed in the intervention.

Based on the findings, CLASP-A will be revised, with the objective of creating a flexible protocol in which emphasis can be shifted based on the presenting problems of the patient/family, and strategies can be selected to accommodate the developmental stage of the patient. CLASP-A is innovative in that it targets the highest risk adolescents during their highest risk period, i.e. transition from inpatient to outpatient care. It is also innovative in employing multiple modalities (in-person sessions and phone calls) that involve both the patient and the parent, thus targeting frequently cited barriers in the treatment of adolescent patients. The availability of a low-cost, easily implemented, adjunctive intervention that successfully reduces the rate of suicide attempts in adolescents could improve quality of life and productivity on both individual and societal levels.

ELIGIBILITY:
Inclusion Criteria:

* Admission to an inpatient unit due to suicide risk
* English speaking

Exclusion Criteria:

* Active psychosis
* Cognitive Disability

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2012-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Yen, Ph.D., Principal Investigator — Brown University
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Please contact PI for data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adolescent Psychiatric Inpatient Unit
Period: Overall Study
Arm/Group | CLASP-A Intervention | Treatment as Usual
Started | 25 | 25
Completed | 19 | 23
Not Completed | 6 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CLASP-A Intervention | Treatment as Usual | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.96 (1.21) | 15.52 (1.42) | 15.74 (1.32)
Sex/Gender, Customized [Number; unit: participants]
  Male | 3 | 6 | 9
  Female | 21 | 19 | 40
  Other | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 15 | 19 | 34
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Repoorted a Suicide Event
Description: A suicide event is either a suicide attempts (actual, aborted, interrupted), or emergency interventions to intercede an attempt.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | CLASP-A Intervention | Treatment as Usual
Number analyzed (Participants) | 19 | 23
participants | 8 | 8
Statistical Analysis 1: Comparison: CLASP-A Intervention vs Treatment as Usual; Test type: Superiority or Other; p = .87, Chi-squared

ADVERSE EVENTS:
Arm/Group | CLASP-A Intervention | Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 11/19 | 9/23
Other Adverse Events (participants affected / at risk) | 0/19 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CLASP-A Intervention (N=19) | Treatment as Usual (N=23)
Suicide attempt (Psychiatric disorders) | 4 (4) | 3 (4) — Non lethal suicide attempts and subsequent psychiatric hospitalization
Hospitalization for suicidal ideation (Psychiatric disorders) | 3 (7) | 6 (9)
ED visit for suicidal ideation (Psychiatric disorders) | 2 (2) | 0 (0)
ED for drug overdose (Psychiatric disorders) | 1 (1) | 0 (0)
ED for medical evaluation (e.g. frostbite) (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Legal Issues (Social circumstances) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No